CLINICAL TRIAL: NCT05186844
Title: Posttraumatic Stress Disorder in Parents and Children After Discharge From the Pediatric Intensive Care Unit
Acronym: PTSD
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayşegül Karaca, Nurse, Eskisehir Osmangazi University
Other Study IDs: Study1; Ayfer Açıkgöz (Other: Eskisehir OU)
Record Dates: First submitted 2021-10-15; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Posttraumatic Stress Disorder; Parents; Children, Only
Keywords: child, intensive care, parent, PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — The research was conducted as a survey study only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: survey application — Scales and questionnaires were applied to children and their parents according to age groups.

SUMMARY:
Background: If disorders that occur immediately after a trauma are not treated, they may become chronic and turn into severe health problems.

Objectives: This study was conducted with children who had spent time in an intensive care unit and their parents to examine the development of posttraumatic stress disorder (PTSD) in both children and parents.

Methods: The study was a cross-sectional study. A total of 110 children, 98 mothers and 80 fathers were included in the study.

DETAILED DESCRIPTION:
Background: If disorders that occur immediately after a trauma are not treated, they may become chronic and turn into severe health problems.

Objectives: This study was conducted with children who had spent time in an intensive care unit and their parents to examine the development of posttraumatic stress disorder (PTSD) in both children and parents.

Methods: The research was carried out in the intensive care unit of a children's hospital in Turkey. Children between the ages of 8-12 who had spent time in the PICU over the period January 1 - March 1, 2019, who had been discharged from the PICU or transferred into another unit during this time, and who met the research criteria were included in the study. Between these dates, the total number of children discharged from intensive care or transferred into another unit was 166. Of these children, 138 were between the ages of 8-12. During this period, three children who died, two children whose general condition meant they were unable to participate in the study, and 23 children for whom parental consent could not be obtained were excluded from the study. The study was ultimately completed with 110 children. In addition, the parents of the children in the sample group (98 mothers and 80 fathers) who were alive, reachable, and who agreed to participate were included in the study.

Results: A total of 110 children, 98 mothers and 80 fathers who agreed to participate in the study, met the sample selection criteria, and were available throughout were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* The child was between 8-12 years old,
* The child had an accompanying adult present,
* The child was conscious and/or able to communicate verbally,
* The child did not have any intellectual disability,
* There were no challenges in communicating with the family and/or the child (i.e., they spoke Turkish, were able to communicate),
* The child's stay at the PICU was no longer than 29 days,
* The child and their family volunteered to participate in the study.

Exclusion Criteria:

* All participants who do not meet the inclusion criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In the power analysis conducted using the G*power 3.0.10 program and an alpha=0.05 margin of error, the power of the study was 85% for 110 children, 93.3% for the 98 mothers and 81.5% for the 80 fathers.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
application of the post-traumatic stress disorder scale | on day 0-3 of discharge
  post traumatic stress disorder scale applied to children
application of the post-traumatic stress disorder scale | on day 0-3 of discharge
  post traumatic stress disorder scale applied to parents

SECONDARY OUTCOMES:
application of the post-traumatic stress disorder scale | on day 30-40 of discharge
  post traumatic stress disorder scale applied to children

OTHER OUTCOMES:
application of the post-traumatic stress disorder scale | on day 30-40 of discharge
  post traumatic stress disorder scale applied to parents

CONTACTS AND LOCATIONS:
Overall Officials: ayşegül karaca, Principal Investigator — aysegulkaraca_88@hotmail.com
Locations (1):
- Aysegul, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Cannot be shared because it is in the publishing phase.